CLINICAL TRIAL: NCT06260852
Title: Identification of Minimum Focal Points in Vision Curve Formation After Pseudophakic Presbyopia Surgery
Brief Title: Identification of Minimum Focal Points in Vision Curve Formation
Status: Recruiting | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES20/Th8/23-11-2023
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Presbyopia; Pseudophakia; Cataract; Refractive Errors
Keywords: pseudophakic presbyopic correction; premium monovision; trifocal diffractive intraocular lenses; extended depth of field intraocular lenses
MeSH Terms: conditions — Presbyopia; Pseudophakia; Cataract; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premium presbyopia surgery: Participants that underwent uncomplicated pseudophakic presbyopia correction with bilateral premium intraocular lenses (IOL) implantation
  Interventions: Diagnostic Test: Diagnostic Test: Visual Acuity Assessment

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: Visual Acuity Assessment — Uncorrected visual acuity for nine distances (25, 28, 33, 40, 50, 60, 100, 200, 300 cm) examination via a Democritus Digital Acuity & Reading Test (DDART).

SUMMARY:
The primary objective of this study is to identify how many focal points and at which distances are necessary for reliable visual curve formation and area of the curve (AoC) calculation using mathematical models and comparing the results to measurements acquired from participants that underwent uncomplicated pseudophakic presbyopia surgery.

DETAILED DESCRIPTION:
This is a prospective, non-inferiority trial. 80 participants that underwent uncomplicated pseudophakic presbyopia surgery with bilateral premium intraocular lenses (IOL) implantation will be recruited, and their postoperative Visual Curves (VAC) will be evaluated for nine distances (25, 28, 33, 40, 50, 60, 100, 200, 300 cm). Then, using polynomial and spline interpolation methods on the measured data, the aim is to generate a unique polynomial of degree ninc -1 that satisfies all data points.

ELIGIBILITY:
Inclusion Criteria:

* age over 40,
* previous bilateral premium cataract surgery,
* best corrected visual acuity (BCVA) < 0,2 logMAR

Exclusion Criteria:

* taking topical medication to reduce intraocular pressure (IOP),
* macular diseases,
* corneal diseases,
* inability to understand the procedure,
* postoperative astigmatism >1.50 diopters,
* postoperative clouding of the posterior capsule

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants that underwent uncomplicated pseudophakic presbyopia correction with bilateral premium intraocular lenses (IOL) implantation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Visual curves interpolation | 6 months
  Visual curves interpolation after visual acuity assessment in 9 focal points
Area of the curve (AOC) assessment | 6 months
  Calculation of the AOC after visual curve interpolation
Visual acuity assessment | 6 months
  Visual acuity assessment in 9 focal points using DDART chart

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Democritus University of Thrace
Locations (1):
- Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece